CLINICAL TRIAL: NCT01751464
Title: A WrapAround Case Management Program for Youth Injured by Violence: A Feasibility Study
Brief Title: A WrapAround Case Management Program for Youth Injured by Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Carolyn Snider, Assistant Professor, Department of Emergency Medicine, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2012:133
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Intentional Injury
Keywords: youth; violence; injury; emergency department; intervention
MeSH Terms: conditions — Wounds and Injuries; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WrapAround Care (Experimental)
  Interventions: Behavioral: WrapAround Case Management

INTERVENTIONS:
Behavioral: WrapAround Case Management — Youth Injured by Violence will be paired with a support worker who has extensive experience working with youth affected by violence.It is important to note that the wraparound concept involves individualized care planning and management. As such, the specific care plan will be different for each participant. Through early intensive meetings, they will develop a mentoring relationship. They will work with the youth to develop a support team, which may include family, teachers, child welfare workers and truly anyone the youth has decided can help them in their path to making positive choices.

SUMMARY:
This is a feasibility study of a WrapAround Case Management Program for Youth Injured by Violence. Youth (aged 10-24) who have been injured by violence and visit the emergency department will be offered a support worker who will provide WrapAround Case Management. This study is designed to assess the feasibility of recruitment, enrollment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10 - 24 and
2. Presentation to an ED or trauma floor with an injury caused by violence (defined as an injury inflicted by someone else and one of a gunshot wound, stab wound, injury due to blunt object, or injury due to bodily force).

Exclusion Criteria:

1. Unable to consent due to language or brain injury,
2. Sexual assault,
3. Child Abuse
4. Self-Inflicted Injury,
5. Subject is under arrest or
6. Non-resident of Winnipeg.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To estimate the recruitment rate of an ED referral program for injured youth | 6 months
  We will evaluate the proportion of eligible patients who are identified for enrolment and any biases in subject identification

SECONDARY OUTCOMES:
To identify barriers to participation in a hospital-based case management program | 6 months
To determine the average number of contacts and amount of time required per participant | 6 months
To estimate the rates of follow-up among those successfully recruited | 6 months
To determine the most appropriate way to notify the case manager of an eligible participant | 6 months
To determine the most successful enrollment strategy for retention of participants | 6 months
To determine level of engagement between the case manager and youth | 6 months
To determine the most appropriate method of follow-up | 6 months
To determine the impact in violence-related attitudes and behaviours among participants | 6 months
To determine the impact on recurrent intentional injury amongst participants | 6 months
To determine the impact on modifiable risk factors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn E Snider, MD MPH, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Health Sciences Centre, Winnipeg, Manitoba, Canada